CLINICAL TRIAL: NCT03708250
Title: PilBouTox® Project: Prospective and Descriptive Study About Button Battery Poisoning Performed on Data Collected by French Poison Control Centres (PCC)
Brief Title: PilBouTox® Project: Button Battery Poisoning From Data Collected by French Poison Control Centres
Acronym: PILBOUTOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/54
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Button Battery Poisoning
Keywords: button battery; intoxication; oesophageal necrosis; Poison Control Centre; Poisoning
MeSH Terms: conditions — Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Button batteries are found in all householders and can be responsible for poisoning, in particular in children. Unexpected complications and death in children who have ingested button battery have been published for over twenty years in medical literature. There are many questions related to the treatment that remain unanswered, because some data are missing in previously published studies. The main objective of this study is to precisely describe poisoning cases by button battery in order to propose a better management

DETAILED DESCRIPTION:
Button batteries are found in all householders and can be responsible for poisoning, in particular in children. Unexpected complications and death in children who have ingested button battery have been published for over twenty years in medical literature. The most serious cases are those related to the ingestion of button cells, especially in children, when the battery gets stuck in the esophagus. Poison control centres, as well as addictovigilance centres, are regularly called upon for serious poisoning resulting in hospitalization, for which precisely description is most often missing or difficult to obtain and limits the efficiency of the management of these poisonings. So there are many questions related to the treatment that remain unanswered, because some data are missing in previously published studies. For example, in many cases, there is a lack of detail of initial symptoms, delays between symptoms and completion of further tests, follow-ups… A prospective and descriptive study about button battery poisoning performed on data collected by French PCC will be conducted between the 1st June of 2016 and the 31 May of 2018: any call in a PCC that occurred during the period studied and concerning an exposure to a button cell regardless of the route of exposure, the age of the patient, and its symptomatology will be included. The following data will be taken : severe complication, need for surgery, length of hospital stay, death, risk factors concerning the battery (size, voltage), abnormalities at the first fibroscopy.

ELIGIBILITY:
Inclusion Criteria:

Any call that occurred during the period studied in a Poison Control Centre and concerning an exposure to a button cell regardless of the route of exposure, the age of the patient, and its symptomatology.

Exclusion Criteria:

Animal cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone who calls for exposure to a button cell regardless of the route of exposure, the age of the patient, and its symptomatology.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
occurrence of a serious complication | Baseline
  occurrence of a serious complication

SECONDARY OUTCOMES:
Need for surgery | baseline
  Need for surgery
Length of hospital stay | baseline
  Length of hospital stay
Death | baseline
  Death
Battery Size | baseline
  Battery Size
Battery Voltage | baseline
  Battery Voltage
Presence of Lying | baseline
  Presence of Lying
Length of Insertion | baseline
  Length of Insertion
Abnormalities at First Fibroscopy | baseline
  Abnormalities at First Fibroscopy

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Centre Anti Poison, Angers
  - Centre Anti Poison, Lille
  - Centre Anti Poison, Lyon
  - Centre Anti Poison, Marseille
  - Centre Anti Poison, Nancy
  - Centre Anti Poison, Paris
  - Centre Anti Poison, Strasbourg
  - Centre Anti Poison, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Labadie M, Vaucel JA, Courtois A, Nisse P, Legeay M, Medernach C, Patat AM, Von Fabeck K, Gallart JC; French PCC Research Group; Tournoud C, Puskarczyk E. Button Battery Ingestion in Children (PilBouTox(R)): A Prospective Study Describing the Clinical Course and Identifying Factors Related to Esophageal Impaction or Severe Cases. Dysphagia. 2023 Feb;38(1):446-456. doi: 10.1007/s00455-022-10485-7. Epub 2022 Jul 16. PMID 35841456